CLINICAL TRIAL: NCT06190470
Title: Effects of Marijuana on Neuropathic Pain and Spasticity in Spinal Cord Injury Patients
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Nuttaset Manimmanakorn, Rehabilitation Medicine Department Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: HE651146
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Spinal Cord Injury
Keywords: Cannabis; Marijuana; Spinal cord injury; Pain; Spasticity
MeSH Terms: conditions — Spinal Cord Injuries; Marijuana Abuse; Pain; Muscle Spasticity | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The participants will receive cannabis product for 2 weeks. The participants will receive the cannabis product (THC 30mg / 1 ml) manufactured by Faculty of pharmaceutical science KhonKaen University. The participants will gradually increase using the product starting from 1 drop (1.5 mg THC) per day sublingually and can increase using not more than 1 drop per day, until pain or spasticity can be controlled.
  Interventions: Drug: Cannabis
- Placebo group (Placebo Comparator): The participants will receive placebo product manufactured by Faculty of Pharmaceutical Science KhonKaen University for 2 weeks. The participants will gradually increase using the product starting from 1 drop per day sublingually and can increase using not more than 1 drop per day,
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabis — Cannabis product is from the extraction of the powdered, dried and mature pistillate inflorescences of Cannabis sativa L. containing THC 30mg/ml.
  Other Names: Marijuana
  Arms: Experimental group
Drug: Placebo — Placebo is similar to Cannabis product but do not contain THC.
  Other Names: Control/ No cannabis
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to compare effects of marijuana or cannabis on neuropathic pain and spasticity in spinal cord injury patients. The main question is: Does the cannabis product from KhonKaen University reduce neuropathic pain and spasticity in spinal cord injury patients? The research design is a crossover study. The participants will be randomly into 2 groups: group 1 and group 2. The participants received either cannabis or placebo for 2 weeks. After completing treatment, participants were swapped to the other group for 2 weeks, a wash-out period is 2 weeks. The outcome measurements are pain and spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury more than 6 months
* Neuropathic pain
* Pain score > 3
* Do not response to standard medical treatment
* Given inform consent

Exclusion Criteria:

* Allergy to cannabis
* Unstable cardiovascular and pulmonary diseases
* Chronic kidney and liver diseases
* Psychological disease
* Pregnancy or breastfeeding

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 2 weeks
  Visual analog scale

SECONDARY OUTCOMES:
Spasticity | 2 weeks
  Modified Asworth Score
Activities of daily living | 2 weeks
  to assess functional outcome
Quality of life score | 2 weeks
  WHO Bref Quality of life questionnaire
H-reflex | 2 weeks
  Electrodiagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Nuttaset Manimmanakorn, MD, PhD, Principal Investigator — Rehabilitation Medicine Department, Faculty of Medicine, KhonKaen University
Locations (1):
- Faculty of Medicine Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification.
Supporting Information: Study Protocol, CSR
Time Frame: beginning 3 months and ending 5 years following article published
Access Criteria: Researchers who provide a methodologically sound proposal.